CLINICAL TRIAL: NCT04144712
Title: High Versus Low Dose Caffeine as Respiratory Stimulant in Preterm Infants
Brief Title: Caffeine as Respiratory Stimulant in Preterm Infants
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Eslam Mohammed Ali Mazrou, Principal Investigator, Pediatric Resident, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FWA 000017685
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2019-10

CONDITIONS: Apnea of Prematurity
MeSH Terms: conditions — Apnea | interventions — caffeine citrate

STUDY DESIGN:
Intervention Model Description: The current study will be carried on preterm infants admitted to the Neonatal Intensive Care Unit (NICU), Ain Shams University 80 Patients divided into two groups each group will contain 40 subjects Group sample sizes of 40 and 40 achieve 83% power to detect a difference of -7.0 regarding frequency of apnea attacks between the null hypothesis that both group means are 9.0 and the alternative hypothesis that the mean of group 2 is 16.0 with known group standard deviations of 3.7 and 5.2 and with a significance level (alpha) of 0.05000 using a two-sided Mann-Whitney test assuming that the actual distribution is uniform
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- High Dose arm (Experimental): subjects will receive the high dose of the drug
  Interventions: Drug: Caffeine Citrate
- low dose arm (Active Comparator): subject will receive low dose of the drug
  Interventions: Drug: Caffeine Citrate

INTERVENTIONS:
Drug: Caffeine Citrate — study rate of occurrence of Apnea of Prematurity between the 2 groups

SUMMARY:
comparison between rate of occurance of apnea of prematurity AOP when using high and low dose caffeine

DETAILED DESCRIPTION:
Caffeine is one of the widely used medications in the neonatal care units and in spite of its widespread use in preterm infants, there has been little information about the optimal efficient dose in those patients Caffeine therapy for treatment of apnea of prematurity (AOP) is well established over the past few years, yet the optimal loading and maintenance dose of caffeine in preterm infants is not well-studied AOP is a common complication of preterm birth, which affects more than 80 % of neonates with a birth weight less than 1,000 g. Methylxanthine (MGs), including caffeine and theophylline, are a mainstay in the treatment and prevention of AOP The efficiency of caffeine, as a preferred methylxanthine, to stimulate respiration has been well proven as it has a significant favorable impact on neonatal morbidity as bronchopulmonary dysplasia (BPD) and patent ductus arteriosus (PDA) ligation. Also, the results of previous studies revealed that caffeine enhances respiratory muscle strength and lung function followed by easier weaning of mechanical ventilation in premature infants. Besides, a rapid and sustained increase in diaphragmatic activity and tidal volume was reported in preterm infants followed by caffeine administration Previous studies have shown that caffeine citrate was generally well tolerated by premature neonates in clinical trials and declined the incidence of apnea in this population compared with placebo. Also, caffeine is related to superior outcomes due to its lower toxicity and it is a preferred drug for apnea in preterm infants with respiratory problems. It has also a significant function as a noninvasive respiratory support. It facilitates the transition from invasive to noninvasive support, reduces the duration of positive airway pressure support and decreases the risk of BPD in preterm infants The optimum caffeine dose in preterm infants with AOP has not been well studied as well as heterogeneous reports on the optimal loading and maintenance dose of caffeine in several studies in terms of benefits and risks. Many investigations have been conducted about various dosing regimens in the improvement or prevention of respiratory disorders of premature infants. These dosage regimens, although, have been associated with varying degrees of success The aim of this study is to determine if the use of caffeine in doses higher than the currently standard dose can decrease the frequency of apnea in preterm infants without causing significant side effects

ELIGIBILITY:
Inclusion Criteria:

* • Preterm infants with a gestational age <32 weeks in room air or CPAP (prophylactic).

  * Preterm infants with gestational age 32-34 weeks who exhibited apnea of prematurity within the first 10 days of life in room air or CPAP

Exclusion Criteria:

* • Major congenital malformations.

  * Chromosomal anomalies.
  * Preterm infants on mechanical ventilation.
  * Preterm infants on NIPPV.

Max Age: 10 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
High Versus Low Dose Caffeine as Respiratory Stimulant in Preterm Infants | baseline
  assess occurrence of apnea of prematurity between infants receiving high and low dose caffeine

CONTACTS AND LOCATIONS:
Overall Officials: Yasmin A Farid, MD, Study Director — Pediatric Department Faculty of Medicine Ain shams University; Ola G Badr El-Deen, MD, Study Chair — Pediatric Department Faculty of Medicine Ain shams University
Locations (1):
- Faculty of Medicine ain shams University, Cairo, Egypt

REFERENCES:
- [Background] Faramarzi F, Shiran M, Rafati M, Farhadi R, Salehifar E, Nakhshab M. The efficacy and safety of two different doses of caffeine in respiratory function of preterm infants. Caspian J Intern Med. 2018 Winter;9(1):46-53. doi: 10.22088/cjim.9.1.46. PMID 29387319
- [Background] Schmidt B, Roberts RS, Davis P, Doyle LW, Barrington KJ, Ohlsson A, Solimano A, Tin W; Caffeine for Apnea of Prematurity Trial Group. Caffeine therapy for apnea of prematurity. N Engl J Med. 2006 May 18;354(20):2112-21. doi: 10.1056/NEJMoa054065. PMID 16707748
- [Background] Kraaijenga JV, Hutten GJ, de Jongh FH, van Kaam AH. The Effect of Caffeine on Diaphragmatic Activity and Tidal Volume in Preterm Infants. J Pediatr. 2015 Jul;167(1):70-5. doi: 10.1016/j.jpeds.2015.04.040. Epub 2015 May 15. PMID 25982138
- [Background] Mohammed S, Nour I, Shabaan AE, Shouman B, Abdel-Hady H, Nasef N. High versus low-dose caffeine for apnea of prematurity: a randomized controlled trial. Eur J Pediatr. 2015 Jul;174(7):949-56. doi: 10.1007/s00431-015-2494-8. Epub 2015 Feb 3. PMID 25644724
- [Background] Zhao Y, Tian X, Liu G. [Clinical effectiveness of different doses of caffeine for primary apnea in preterm infants]. Zhonghua Er Ke Za Zhi. 2016 Jan;54(1):33-6. doi: 10.3760/cma.j.issn.0578-1310.2016.01.008. Chinese. PMID 26791921